CLINICAL TRIAL: NCT05729932
Title: Cannabis Modulation of Outcomes Related to Opioid Use Disorder: Opioid Withdrawal, Abuse Potential and Safety
Brief Title: Cannabis and Opioid Use Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Shanna Babalonis, PhD, Principal Investigator, University of Kentucky
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 75562-20242; 1R01DA054347 (NIH)
Record Dates: First submitted 2023-01-13; First posted 2023-02-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Opioid Agonist (Experimental): Participants will receive non-therapeutic, experimental doses of an opioid agonist or placebo. Active opioid agonist/placebo will be administered once per session and will be administered intransally (snorting).
  Interventions: Drug: Inhaled vaporized cannabis; Drug: Intransal opioid
- Vaporized cannabis (Experimental): Participants will receive non-therapeutic, experimental doses of active or placebo vaporized cannabis. Active cannabis/placebo will be administered once per session and will be administered via a vaporizer.
  Interventions: Drug: Inhaled vaporized cannabis; Drug: Intransal opioid

INTERVENTIONS:
Drug: Inhaled vaporized cannabis — Double-blind cannabis and placebo doses, administered through vaporizer
Drug: Intransal opioid — Double-blind opioid and placebo doses, administered intranasal route

SUMMARY:
This study plans to enroll participants with opioid use disorder who are not currently seeking treatment to assess the effects of cannabis on opioid withdrawal and other related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid use disorder

Exclusion Criteria:

* Current medical conditions that require medical management

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline - Opioid Withdrawal Severity - Visual Analog Scale (VAS) | Change from baseline
  Subjective ratings of opioid withdrawal severity on visual analog scale (scale 0-100; 0 = not at all, 100 = extremely)

SECONDARY OUTCOMES:
Change from Baseline - Opioid Drug Liking - Visual Analog Scale (VAS) | Change from baseline
  Subjective ratings of drug liking on visual analog scale (scale 0-100, 0 = not at all, 100 = extremely)
Change from Baseline - Respiration | Change from baseline
  Physiological monitoring of respiration rate (breaths per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Shanna Babalonis, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Center on Drug and Alcohol Research, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No